CLINICAL TRIAL: NCT00003909
Title: A Phase I Study of Motexafin Gadolinium (Xcytrin, NSC 695238) and Involved Field Radiation Therapy for Intrinsic Pontine Glioma of Childhood
Brief Title: Motexafin Gadolinium Plus Radiation Therapy in Treating Children With Newly Diagnosed Brain Stem Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01845; COG-A09712; U01CA097452 (NIH); CDR0000067087 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Untreated Childhood Brain Stem Glioma
MeSH Terms: interventions — motexafin gadolinium; Radiotherapy; Radiation

ARMS (1):
- Arm I (Experimental): Approximately 2-5 hours before radiotherapy, patients receive motexafin gadolinium IV over 5 minutes. Patients undergo radiotherapy 5 days a week for 6 weeks.
  Interventions: Drug: motexafin gadolinium; Radiation: radiation therapy; Other: pharmacological study

INTERVENTIONS:
Drug: motexafin gadolinium — Given IV
  Other Names: gadolinium texaphyrin; Gd (III) Texaphryin; Gd-Tex; PCI-0120; Xcytrin
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: pharmacological study — Correlatives studies
  Other Names: pharmacological studies

SUMMARY:
Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as motexafin gadolinium may make the tumor cells more sensitive to radiation therapy. Phase I trial to study the effectiveness of motexafin gadolinium plus radiation therapy in treating children who have newly diagnosed brain stem glioma

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and schedule of motexafin gadolinium administered prior to radiotherapy in children with newly diagnosed diffuse intrinsic pontine glioma.

II. Determine the toxic effects of this drug given at the MTD in these patients.

III. Determine the intratumor and brain distribution of this drug by magnetic resonance imaging (MRI) in these patients.

OUTLINE: This is a dose-escalation study of motexafin gadolinium.

Approximately 2-5 hours before radiotherapy, patients receive motexafin gadolinium IV over 5 minutes. Patients undergo radiotherapy 5 days a week for 6 weeks.

Cohorts of 3-6 patients receive escalating doses of motexafin gadolinium until the MTD is determined. The first cohort receives motexafin gadolinium 5 days a week for 3 weeks; the second cohort receives motexafin gadolinium 3 days a week for 6 weeks; and subsequent cohorts receive motexafin gadolinium 5 days a week for 6 weeks. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for up to 3 years.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and radiographically (MRI) proven newly diagnosed diffuse intrinsic brainstem glioma

  * Greater than 50% intra-axial involvement of the pons, pons and medulla, pons and midbrain, or entire brainstem
  * Contiguous involvement of the thalamus or upper cervical cord allowed
* Performance status - ECOG 0-2
* More than 2 months
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL (transfusion allowed)
* No glucose 6 phosphate dehydrogenase deficiency
* Bilirubin no greater than 1.5 times normal
* SGOT or SGPT less than 1.5 times normal
* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent immunomodulating agents
* No other concurrent chemotherapy
* Concurrent corticosteroid therapy allowed for increased intracranial pressure only
* No prior cranial radiotherapy
* No prior motexafin gadolinium
* No other concurrent experimental agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 1999-08; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose at which fewer than one-third of patients experience DLT assessed using CTC version 2.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minesh Mehta, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States